CLINICAL TRIAL: NCT00099606
Title: A Phase I Dose-Escalation Study of BMS-354825 in Patients With Refractory Solid Tumors
Brief Title: Phase I (PH I) Mad Refractory Solid Tumor Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA180-003
Record Dates: First submitted 2004-12-17; First posted 2004-12-20 (Estimated); Last update posted 2011-04-19 (Estimated); Status verified 2011-04

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — Dasatinib

ARMS (1):
- A1 (Experimental)
  Interventions: Drug: Dasatinib

INTERVENTIONS:
Drug: Dasatinib — Tablets, Oral, Dose Finding Study - Range was 35 mg BID, 5 days on/2 days off - 120 mg BID Continuous Daily Dosing, Once daily, Patients remained on study until treatment discontinuation due to unacceptable toxicity, disease progression or death.
  Other Names: Sprycel

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics, effect of food, and continue exploratory research of BMS-354825 in patients with solid tumors not responding to standard treatment, or for which no effective standard treatment exists.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Available for protocol-required follow-up
* ECOG performance status score 0 - 1 (See Appendix 1)
* Histologic or cytologic diagnosis of a primary solid (i.e., non-hematologic) malignancy
* Evidence (radiographic or tissue confirmation) that the disease is metastatic
* Metastatic disease which has progressed on or following currently available standard therapies or for which no standard therapy exists. (Prior adjuvant or neoadjuvant therapy is permitted. Prior investigational agents are permitted);
* Measurable or non-measurable disease as defined in Section 3.3.2.1
* Adequate bone marrow function defined as:
* absolute neutrophil count (neutrophil and bands) >=2,000 cells/mm3
* platelet count >=125,000 cells/mm3
* hemoglobin >=9.0 g/dl
* Adequate hepatic function defined as:
* total bilirubin <=1.5 times the institutional upper limit of normal,
* alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <=2.0 times the institutional upper limit of normal
* Adequate renal function defined as:
* serum creatinine <=1.5 times the institutional upper normal limit
* Serum potassium and magnesium levels within institutional normal limits. Total serum calcium or ionized calcium level must be greater than or equal to the lower limit of normal. Patients with low potassium and magnesium levels may be repleted to allow for protocol entry.
* CD4+ T-cell counts of >=the institutional lower limit of normal.
* Prior chemo-, radio-, hormonal or immunotherapy are allowed. Patients must have recovered from toxicity due to prior therapy i.e., toxicity has resolved to baseline or is deemed irreversible. At least 4 weeks must have elapsed since the last chemotherapy (6 weeks for nitrosoureas, mitomycin-C, and liposomal doxorubicin), immunotherapy or radiotherapy and the beginning of protocol therapy. At least 2 weeks must have elapsed since last hormonal therapy or exposure to any other "targeted" kinase inhibitor (e.g., imatinib mesylate).
* Bleeding time <=upper limit of institutional normal or platelet aggregometry result within the institutional normal limits
* Men and women, ages 18 and older. Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for a period of at least 1 month prior and at least 3 months after the study in such a manner that the risk of pregnancy is minimized.

WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation or bilateral oophorectomy) or is not postmenopausal [defined as amenorrhea >=12 consecutive months; or women on hormone replacement therapy (HRT) with documented serum follicle stimulating hormone (FSH) level >35 mIU/mL]. Even women who are using oral, implanted or injectable contraceptive hormones or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy or practicing abstinence or where partner is sterile (e.g., vasectomy), should be considered to be of child bearing potential.

WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours prior to the start of study medication.

Exclusion Criteria:

* WOCBP who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period including the period from one month prior to starting study medication and for a period of at least 3 months after the study.
* WOCBP using a prohibited contraceptive method.
* Women who are pregnant or breastfeeding.
* Women with a positive pregnancy test on enrollment or prior to study drug administration.
* Men who are unwilling or unable to use an acceptable method of birth control for the entire study period and for at least 3 months after completion of study medication if their sexual partners are WOCBP.
* Received extensive prior radiation therapy to the bone marrow. Generally, patients should have radiation to <=25% of bone marrow-containing skeleton (see Appendix 2).
* Known brain metastasis. Patients with symptoms of brain metastasis are not eligible unless brain metastasis are ruled out by CT or MRI.
* A serious uncontrolled medical disorder or active infection which would impair the ability of the patient to receive protocol therapy.
* Uncontrolled or significant cardiovascular disease, including:
* A myocardial infarction within 12 months
* Uncontrolled angina within 6 months
* Congestive heart failure within 6 months
* Diagnosed or suspected congenital long QT syndrome
* Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or torsade de pointes). Any patient with a history of any arrhythmia should be discussed with the BMS Medical Monitor prior to entry into the study.
* Prolonged QTc interval on pre-entry electrocardiogram (> 450 msec)
* Any history of second or third degree heart block (may be eligible if currently have a pacemaker)
* Heart rate < 50 / minute on pre-entry electrocardiogram
* Uncontrolled hypertension.
* Dementia or altered mental status that would prohibit the understanding or rendering of informed consent;
* History of significant bleeding disorder including:
* Diagnosed congenital bleeding disorders (e.g., von Willebrand's disease)
* Diagnosed acquired bleeding disorder within one year (e.g., acquired anti-factor VIII antibodies)
* Documented major bleeding episode from the GI tract within 6 months unless no longer at significant risk due to surgical intervention
* Vasculitis.
* Received investigational agents within 4 weeks prior to the start of protocol therapy.
* Patients currently taking drugs that are generally accepted to have a risk of causing Torsades de Pointes including:
* Class IA antiarrhythmic agents (quinidine, procainamide, disopyramide, mexiletine)
* Class III antiarrhythmic agents ( amiodarone, sotalol, ibutilide, dofetilide)
* Macrolide antibiotics (erythromycins, clarithromycin)
* Antipsychotics (chlorpromazine, haloperidol, mesoridazine, thioridazine, pimozide)
* Tricyclic antidepressants
* Miscellaneous (cisapride, bepridil, inapsine, methadone, arsenic). Patients who have discontinued any of these medications must have a wash-out period of at least 5 days or at least 5 half-lives of the drug (whichever is greater) prior to the first dose of BMS-354825.
* Patients taking medications that inhibit platelet function (e.g., aspirin, dipyridamole, epoprostenol, eptifibatide, clopidogrel, cilostazol, abciximab, ticlopidine, and any non-steroidal anti-inflammatory drug) or anticoagulants (warfarin, heparin/low molecular weight heparin [e.g., danaparoid, dalteparin, tinzaparin, enoxaparin]). Patients who have discontinued aspirin must have a wash-out period of at least 7 days for low-dose aspirin (<=325 mg/day) or 14 days for higher-dose aspirin (> 325 mg/day) prior to the first dose of BMS-354825. Patients who have discontinued other antiplatelet or anticoagulant medications must have a wash-out period of at least 5 days or at least 5 half lives of the drug (whichever is greater) prior to the first dose of BMS-354825.
* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious disease) illness must not be enrolled into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2004-07; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Phase I-Dose Escalation to Determine MTD, Safety

SECONDARY OUTCOMES:
Pharmocokinetics

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (3):
- United States (2):
  - Local Institution, Boston, Massachusetts
  - Local Institution, Detroit, Michigan
- Local Institution, Glasgow, Strathclyde, United Kingdom

REFERENCES:
- [Background] Demetri GD, Lo Russo P, MacPherson IR, Wang D, Morgan JA, Brunton VG, Paliwal P, Agrawal S, Voi M, Evans TR. Phase I dose-escalation and pharmacokinetic study of dasatinib in patients with advanced solid tumors. Clin Cancer Res. 2009 Oct 1;15(19):6232-40. doi: 10.1158/1078-0432.CCR-09-0224. Epub 2009 Sep 29. PMID 19789325